CLINICAL TRIAL: NCT00027417
Title: Triostat in Children During CardioPulmonary Bypass (CPB)
Brief Title: Study of Triostat in Infants During Heart Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Michael Portman (Other)
Responsible Party: Sponsor-Investigator, Michael Portman, Cardiologist, Seattle Children's Hospital
Organization: Seattle Children's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FD-R-1971-01; FD-R-001971-01
Record Dates: First submitted 2001-12-05; First posted 2001-12-07 (Estimated); Last update posted 2013-08-05 (Estimated); Status verified 2013-08

CONDITIONS: Heart Defects, Congenital
Keywords: Congenital heart defects; Hypoplastic left heart syndrome; Complete atrioventricular canal defect; Triostat; Cardiac surgery
MeSH Terms: conditions — Heart Defects, Congenital; Hypoplastic Left Heart Syndrome; Endocardial Cushion Defects | interventions — Triiodothyronine; Cardiopulmonary Bypass; Cardiac Surgical Procedures

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Liothyronine Sodium/Triiodothyronine (Active Comparator): bolus administration of Liothyronine Sodium/Triiodothyronine (Triostat) immediately prior to CPB institution and after removal of aortic cross clamp, followed by repeated boluses, will be safe and will result in significant improvements in postoperative and clinical outcome parameters and cardiac contractile function.
  Interventions: Drug: Liothyronine sodium/triiodothyronine; Procedure: Cardiopulmonary bypass and cardiac surgery
- Placebo (Placebo Comparator): bolus administration of Placebo immediately prior to CPB institution and after removal of aortic cross clamp, followed by repeated boluses
  Interventions: Drug: Liothyronine sodium/triiodothyronine; Procedure: Cardiopulmonary bypass and cardiac surgery

INTERVENTIONS:
Drug: Liothyronine sodium/triiodothyronine
Procedure: Cardiopulmonary bypass and cardiac surgery

SUMMARY:
This is a study to determine the safety and efficacy of liothyronine sodium/triiodothyronine (Triostat), a synthetic thyroid hormone, when given to infants with congenital heart disease during cardiopulmonary bypass surgery.

DETAILED DESCRIPTION:
Patients will be randomized to receive study drug or placebo and randomization will occur stratified to each diagnostic category. All patients undergo preoperative echocardiograms to provide preoperative cardiac function data. The study drug or placebo will be provided in the operating room as an iv bolus just prior to cardiopulmonary bypass and as a bolus delivered on release of the aortic cross-clamp. This will be followed by iv for 12 hours. Operative data will be collected including CPB time, aortic cross-clamp time, length and degree of hypothermia. These data will be extracted from the anesthesia record.

ELIGIBILITY:
Inclusion criteria:

Diagnosis of one of the following:

* Ventricular septal defect (VSD)
* Infant coarctation of the aorta
* Transposition of the great arteries
* Tetralogy of Fallot
* Complete atrioventricular canal defect
* Hypoplastic left heart, including patients who undergo a Norwood type procedure for aortic or mitral atresia

Patient must be scheduled for surgery.

Exclusion criteria:

* Certain additional defects and/or requirement for additional surgery.

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 195 (Actual)
Dates: Start 2001-04; Primary Completion 2007-08 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
duration of mechanical ventilation after cardiopulmonary bypass. | 0 to 72 hours
  Reducing the length of ventilatory support minimizes other postoperative complications, which can contribute to morbidity.

SECONDARY OUTCOMES:
Assess other parameters | 0 to 72 hrs
  * Need for mechanic circulatory support, fluid balance (intake and output); urine output
  * Echocardiographic measures to include end-systolic wall stress/fractional shortening ratio
  * Myocardial performance index (Doppler derived), cardiac index (Doppler derived)
  * Heart rate, blood pressure and central venous pressure
  * Free and total T3 levels
  * Others: All medications including inotropic agents will be recorded with respect to time initiated, terminated, and dosage will be recorded for exploratory analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Portman, MD, Principal Investigator — Seattle Childrens Hospital
Locations (1):
- Children's Hospital and Regional Medical Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Portman MA, Slee A, Olson AK, Cohen G, Karl T, Tong E, Hastings L, Patel H, Reinhartz O, Mott AR, Mainwaring R, Linam J, Danzi S; TRICC Investigators. Triiodothyronine Supplementation in Infants and Children Undergoing Cardiopulmonary Bypass (TRICC): a multicenter placebo-controlled randomized trial: age analysis. Circulation. 2010 Sep 14;122(11 Suppl):S224-33. doi: 10.1161/CIRCULATIONAHA.109.926394. PMID 20837917